CLINICAL TRIAL: NCT01098903
Title: Predictive Value of Drug Elimination Gene Polymorphisms on Clearance and Dose Adjustment of Sunitinib (Sutent, SU11248) in Patients With Cancer
Brief Title: Predictive Value of Drug Elimination Gene Polymorphisms on Clearance and Dose Adjustment of Sunitinib in Cancer Patients
Acronym: CLEARSUN
Status: Completed | Type: Observational
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Collaborators: Erasmus Medical Center (Other); South West Sydney Local Health District (Other)
Responsible Party: Principal Investigator, Heinz-Josef Klumpen, md, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Other Study IDs: HGWH0008
Record Dates: First submitted 2010-03-16; First posted 2010-04-05 (Estimated); Last update posted 2012-07-12 (Estimated); Status verified 2012-07

CONDITIONS: Cancer
Keywords: sunitinib; cancer; pharmacogenomics; pharmacokinetics; Patients who have a malignancy and are going to be treated with sunitinib; doseindividualism
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Sunitinib: Patients with a malignancy treated with sunitinib

SUMMARY:
Sunitinib is an anticancer drug, but like most drugs, the effect varies from person to person. This is partly due to a variation in how well each person eradicates the drug from the body. This can lead to toxicity if the drug is eliminated slowly. Just as important is inadvertent underdosing in people who eliminate the drug quickly which may lead to a reduced anti-cancer effect. The investigators group has developed a battery of tests that may measure how an individual clears a drug from their body. The investigators intend to apply these tests to a group of patients taking sunitinib to see whether any test will help predict the level of sunitinib in the body and also the side effects. If a test seems to be promising from this study it may be possible to do a simple test on patients before they receive sunitinib so the best dose is chosen. The tests involve identifying the genes that are involved with drug elimination (CYP3A, ABCB1, ABCG2, OCT1, OATP) as well as directly measuring elimination using marker drugs (midazolam clearance and sestamibi liver clearance).

ELIGIBILITY:
Inclusion Criteria:

* Age >18
* A malignancy treated with single agent sunitinib
* ECOG 0, 1 or 2 at time of study accruement
* Any stable dose of therapy with sunitinib (defined as no dose change within 3 weeks prior to blood collection for pharmacokinetics)
* Adequate liver and renal function defined as serum bilirubin concentration less than 2 x ULN, AST and ALT less than 2.5 x ULN, serum creatinine concentration less than 2 x ULN
* No known primary liver disease and no other severe or uncontrolled concurrent medical condition within the first 3 months of treatment with sunitinib.
* Patients who have participated on other clinical studies of sunitinib will be suitable for this study.
* Signed informed consent
* Patients must not have Class ¾ cardiac problems as defined by the New York Heart Association criteria or any other severe or uncontrolled concurrent medical disease.
* Patients must not be pregnant or nursing and must be using an effective contraception method

Exclusion Criteria:

* Patients who are unable to sign informed consent
* Patients unable to give blood
* Patients with known midazolam allergies will not be included
* Patients must not be pregnant or nursing and must be using an effective contraception method
* Patients who had a bone-marrow-transplantation prior to sunitinib treatment
* Patients must not be taking routine systemic corticoid therapy
* Patients must not be taking therapeutic warfarin or warfarin derivates doses as anticoagulation at the time of study tests with an at least 2 weeks warfarin free period of time prior. Patients requiring anticoagulation may use low-molecular weight heparin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a malignancy treated with sunitinib
Sampling Method: Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2009-01; Primary Completion 2011-06 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
To observe the correlation between ABCB1 polymorphisms in Exons 13, 22 and 27 and the clearance of sunitinib at steady state. | 4 weeks
  A blood sample will be drawn on day 1 of any treatment cycle and at steady state of the same cycle (between Day 21 and 28 inclusive)

SECONDARY OUTCOMES:
To determine whether ABCB1 genotype correlates with toxicity-adjusted dose of sunitinib | 3 months
  Toxicity adjustments will be collected within the first 3 months and correlated with the ABCB1 genotypes.
To determine the pharmacokinetics at steady state of the sunitinib treatment. | 4 weeks
  A blood sample will be drawn on day 1 of treatment cycle and at steady state of the same cycle (between Day 21 and 28 inclusive). The time of the blood collection are at day1 and in the 4th week: pre-drug administration then at 4 hours, 8 hours and 24 hours after drug intake.
To examine correlations between ABCB1 genotype and toxicity grade according to CTC criteria. | 3 months
  The toxicity data of the first 3 months of treatment will be collected.
To examine the correlation between genotype haplotype of other drug elimination genes, such as organic anion transporter proteins (OATP) and other biliary efflux proteins such as MRP2, BCRP with sunitinib clearance and toxicity adjusted dose. | 3 months
  Investigations of drugelimination and clearance taken with in the first 4 weeks of the study will be collected as well as the toxicity data and dose adjustments within the first 3 month of treatment.
Correlation of drug elimination phenotype test (sestamibi liver scan and Midazolam clearance) with sunitinib clearance | 4 weeks
  sestamibi liver scan and midazolam clearance test will be performed pre-treatment and at steady state (sometime between day 21-28)of study participation.

CONTACTS AND LOCATIONS:
Locations (3):
- Westmead Hospital, Westmead, New South Wales, Australia
- Netherlands (2):
  - Academic medical center Amsterdam, Amsterdam
  - Erasmus Medical Center, Daniel Den Hoed Cancer Center, Rotterdam